CLINICAL TRIAL: NCT01210001
Title: A Randomised, Double-blind, Placebo-controlled Parallel Group Efficacy and Safety Trial of BI 10773 (10 and 25 mg Administered Orally Once Daily) Over 24 Weeks in Patients With Type 2 Diabetes Mellitus With Insufficient Glycaemic Control Despite a Background Therapy of Pioglitazone Alone or in Combination With Metformin
Brief Title: Efficacy and Safety of Empagliflozin (BI 10773) in Type 2 Diabetes Patients on a Background of Pioglitazone Alone or With Metformin
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1245.19; 2009-016154-40 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — empagliflozin

ARMS (3):
- BI 10773 low dose (Experimental): BI 10773 tablets once daily
  Interventions: Drug: BI 10773; Drug: Placebo
- BI 10773 high dose (Experimental): BI 10773 tablets once daily
  Interventions: Drug: Placebo; Drug: BI 10773
- Placebo (Placebo Comparator): Placebo tablets matching BI 10773
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo tablets matching BI 10773 low dose
  Arms: Placebo
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 low dose
Drug: Placebo — Placebo tablets matching BI 10773 high dose
  Arms: BI 10773 high dose
Drug: Placebo — Placebo tablets matching BI 10773 high dose
  Arms: BI 10773 low dose
Drug: Placebo — Placebo tablets matching BI 10773 high dose
  Arms: Placebo
Drug: BI 10773 — BI 10773 tablets once daily
  Arms: BI 10773 high dose

SUMMARY:
This study will investigate the efficacy and safety of BI 10773 in type 2 diabetic patients in order to provide these data for approval for BI 10773 by regulatory authorities as an antidiabetic agent as add-on therapy to pioglitazone alone or in combination with metformin.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of type 2 diabetes mellitus prior to informed consent.
2. Male and female patients on diet and exercise regimen who are pre-treated with pioglitazone alone or in combination with metformin. The treatment regimen should be unchanged for 12 weeks prior to randomisation.
3. HbA1c of >/= 7.0% and </= 10.0% at Visit 1 (screening).
4. Age >/= 18.
5. BMI </= 45 kg/m2 (Body Mass Index) at Visit 1 (screening).
6. Signed and dated written informed consent by date of Visit 1 in accordance with Good Clinical Practice (GCP) and local legislation.

Exclusion criteria:

1. Uncontrolled hyperglycaemia with a glucose level > 240 mg/dl (> 13.3 mmol/l) after an overnight fast during placebo run-in and confirmed by a second measurement (not on the same day).
2. Any other antidiabetic medication within 12 weeks prior to randomisation, except those defined as the permitted background therapy via inclusion criteria no. 2.
3. Myocardial infarction, stroke or transient ischaemic attack (TIA) within 3 months prior to informed consent.
4. Indication of liver disease, defined by serum levels of either alanine transaminase (ALT/SGPT), aspartate transaminase (AST/SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined during screening or during the placebo run-in period (i.e. at a visit prior to the randomisation visit, Visit 3).
5. Impaired renal function, defined as eGFR (estimated Glomerular Filtration Rate) < 30 ml/min (severe renal impairment, MDRD [Modification of Diet in Renal Disease] formula) as determined during screening or during the placebo run-in period (i.e. at a visit prior to the randomisation visit, Visit 3).
6. Bariatric surgery within the past two years and other gastrointestinal surgeries that induce chronic malabsorption.
7. Medical history of cancer (except for basal cell carcinoma) and/or treatment for cancer within the last 5 years .
8. Blood dyscrasias or any disorders causing haemolysis or unstable red blood cells (e.g. malaria, babesiosis, haemolytic anaemia).
9. Contraindications to pioglitazone according to the local label.
10. Contraindication to pioglitazone and/or metformin (relevant only for those patients who enter the study with both these background therapies) according to the local labels.
11. Treatment with anti-obesity drugs (e.g. sibutramine, orlistat) 3 months prior to informed consent or any other treatment at the time of screening (i.e. surgery, aggressive diet regimen etc.) leading to unstable body weight.
12. Current treatment with systemic steroids at time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent or any other uncontrolled endocrine disorder except T2D.
13. Pre-menopausal women (last menstruation </= 1 year prior to informed consent) who:

    * are nursing or pregnant or
    * are of child bearing potential and are not practicing an acceptable method of birth control, or do not plan to continue using this method throughout the trial and do not agree to submit to periodic pregnancy testing during participation in the trial. Acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence (if acceptable to local authorities), double barrier method and vasectomised partner.
14. Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation or any ongoing condition leading to a decreased compliance to study procedures or study drug intake.
15. Participation in another trial with an investigational drug within 30 days prior to informed consent.
16. Any other clinical condition that would jeopardise patient safety while participating in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 499 (Actual)
Dates: Start 2010-09; Primary Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (68):
- United States (24):
  - 1245.19.10056 Boehringer Ingelheim Investigational Site, Muscle Shoals, Alabama
  - 1245.19.10162 Boehringer Ingelheim Investigational Site, Glendale, Arizona
  - 1245.19.10161 Boehringer Ingelheim Investigational Site, Phoenix, Arizona
  - 1245.19.10046 Boehringer Ingelheim Investigational Site, Tempe, Arizona
  - 1245.19.10070 Boehringer Ingelheim Investigational Site, Irvine, California
  - 1245.19.10047 Boehringer Ingelheim Investigational Site, La Mesa, California
  - 1245.19.10149 Boehringer Ingelheim Investigational Site, Rancho Cucamonga, California
  - 1245.19.10163 Boehringer Ingelheim Investigational Site, Riverside, California
  - 1245.19.10131 Boehringer Ingelheim Investigational Site, West Hills, California
  - 1245.19.10141 Boehringer Ingelheim Investigational Site, Milford, Connecticut
  - 1245.19.10133 Boehringer Ingelheim Investigational Site, Jupiter, Florida
  - 1245.19.10085 Boehringer Ingelheim Investigational Site, Plantation, Florida
  - 1245.19.10077 Boehringer Ingelheim Investigational Site, Perry, Georgia
  - 1245.19.10014 Boehringer Ingelheim Investigational Site, Dubuque, Iowa
  - 1245.19.10160 Boehringer Ingelheim Investigational Site, Essex, Maryland
  - 1245.19.10003 Boehringer Ingelheim Investigational Site, Dearborn, Michigan
  - 1245.19.10059 Boehringer Ingelheim Investigational Site, New Hyde Park, New York
  - 1245.19.10123 Boehringer Ingelheim Investigational Site, Smithtown, New York
  - 1245.19.10071 Boehringer Ingelheim Investigational Site, Asheboro, North Carolina
  - 1245.19.10086 Boehringer Ingelheim Investigational Site, Salisbury, North Carolina
  - 1245.19.10008 Boehringer Ingelheim Investigational Site, Marion, Ohio
  - 1245.19.10033 Boehringer Ingelheim Investigational Site, Chattanooga, Tennessee
  - 1245.19.10112 Boehringer Ingelheim Investigational Site, Memphis, Tennessee
  - 1245.19.10002 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
- Canada (11):
  - 1245.19.20047 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1245.19.20062 Boehringer Ingelheim Investigational Site, Vancouver, British Columbia
  - 1245.19.20012 G.A. Research Associates Ltd., Moncton, New Brunswick
  - 1245.19.20031 Boehringer Ingelheim Investigational Site, St. John's, Newfoundland and Labrador
  - 1245.19.20057 Boehringer Ingelheim Investigational Site, Brampton, Ontario
  - 1245.19.20059 Boehringer Ingelheim Investigational Site, Fort Erie, Ontario
  - 1245.19.20060 Boehringer Ingelheim Investigational Site, London, Ontario
  - 1245.19.20009 Boehringer Ingelheim Investigational Site, Newmarket, Ontario
  - 1245.19.20034 Boehringer Ingelheim Investigational Site, Sarnia, Ontario
  - 1245.19.20058 Boehringer Ingelheim Investigational Site, Saint Romuald, Quebec
  - 1245.19.20041 Boehringer Ingelheim Investigational Site, Saskatoon, Saskatchewan
- Greece (3):
  - 1245.19.30002 Boehringer Ingelheim Investigational Site, Athens
  - 1245.19.30001 Boehringer Ingelheim Investigational Site, Nikaia
  - 1245.19.30004 Boehringer Ingelheim Investigational Site, Thessaloniki
- India (17):
  - 1245.19.91005 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.19.91006 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.19.91008 Boehringer Ingelheim Investigational Site, Bangalore
  - 1245.19.91003 Boehringer Ingelheim Investigational Site, Belagavi
  - 1245.19.91004 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.19.91009 Boehringer Ingelheim Investigational Site, Chennai
  - 1245.19.91001 Boehringer Ingelheim Investigational Site, Coimbatore
  - 1245.19.91015 Boehringer Ingelheim Investigational Site, Kalaburagi
  - 1245.19.91011 Boehringer Ingelheim Investigational Site, Kartanaka
  - 1245.19.91002 Boehringer Ingelheim Investigational Site, Mumbai
  - 1245.19.91007 Boehringer Ingelheim Investigational Site, Mumbai, Maharastra
  - 1245.19.91017 Boehringer Ingelheim Investigational Site, Mysore
  - 1245.19.91010 Boehringer Ingelheim Investigational Site, Nagpur
  - 1245.19.91012 Boehringer Ingelheim Investigational Site, New Delhi
  - 1245.19.91013 Boehringer Ingelheim Investigational Site, Patna
  - 1245.19.91014 Boehringer Ingelheim Investigational Site, Pune
  - 1245.19.91016 Boehringer Ingelheim Investigational Site, Pune
- Philippines (5):
  - 1245.19.63002 Boehringer Ingelheim Investigational Site, Cebu City, N/A, Philippines
  - 1245.19.63003 Boehringer Ingelheim Investigational Site, Davao City, N/A, Philippines
  - 1245.19.63004 Boehringer Ingelheim Investigational Site, Manila, Philippines
  - 1245.19.63005 Boehringer Ingelheim Investigational Site, Pasig City, Philippines
  - 1245.19.63001 Boehringer Ingelheim Investigational Site, San Juan City, Philippines
- Thailand (2):
  - 1245.19.66003 Boehringer Ingelheim Investigational Site, Saimai
  - 1245.19.66004 Boehringer Ingelheim Investigational Site, Udon Thani, Thailand
- Ukraine (6):
  - 1245.19.75002 Boehringer Ingelheim Investigational Site, Dnipro
  - 1245.19.75001 Boehringer Ingelheim Investigational Site, Kharkiv
  - 1245.19.75005 Boehringer Ingelheim Investigational Site, Kiev
  - 1245.19.75006 Boehringer Ingelheim Investigational Site, Lviv
  - 1245.19.75004 Boehringer Ingelheim Investigational Site, Vinnitsa
  - 1245.19.75003 Boehringer Ingelheim Investigational Site, Vinnytsia

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818
- [Derived] Tuttle KR, Levin A, Nangaku M, Kadowaki T, Agarwal R, Hauske SJ, Elsasser A, Ritter I, Steubl D, Wanner C, Wheeler DC. Safety of Empagliflozin in Patients With Type 2 Diabetes and Chronic Kidney Disease: Pooled Analysis of Placebo-Controlled Clinical Trials. Diabetes Care. 2022 Jun 2;45(6):1445-1452. doi: 10.2337/dc21-2034. PMID 35472672
- [Derived] Cherney D, Lund SS, Perkins BA, Groop PH, Cooper ME, Kaspers S, Pfarr E, Woerle HJ, von Eynatten M. The effect of sodium glucose cotransporter 2 inhibition with empagliflozin on microalbuminuria and macroalbuminuria in patients with type 2 diabetes. Diabetologia. 2016 Sep;59(9):1860-70. doi: 10.1007/s00125-016-4008-2. Epub 2016 Jun 17. PMID 27316632
- [Derived] Kovacs CS, Seshiah V, Merker L, Christiansen AV, Roux F, Salsali A, Kim G, Stella P, Woerle HJ, Broedl UC; EMPA-REG EXTEND PIO investigators. Empagliflozin as Add-on Therapy to Pioglitazone With or Without Metformin in Patients With Type 2 Diabetes Mellitus. Clin Ther. 2015 Aug;37(8):1773-88.e1. doi: 10.1016/j.clinthera.2015.05.511. Epub 2015 Jun 29. PMID 26138864

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: A placebo tablet, matching the empagliflozin 10mg and 25mg tablets, taken once daily for 24 weeks
- Empa 10mg: Single oral dose of empagliflozin (empa) 10mg taken once daily for 24 weeks
- Empa 25mg: Single oral dose of empagliflozin (empa) 25mg taken once daily for 24 weeks
Period: Overall Study
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Started | 166 | 165 | 168
Completed | 147 | 154 | 156
Not Completed | 19 | 11 | 12
Not completed — Not treated | 1 | 0 | 0
Not completed — Adverse Event | 4 | 2 | 5
Not completed — Non compliant with protocol | 2 | 2 | 3
Not completed — Lost to Follow-up | 4 | 3 | 2
Not completed — Patient refusal to continue,not due toAE | 6 | 2 | 1
Not completed — Other reason not defined above | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Population: Treated set (TS): all patients treated with at least one dose of randomised study medication
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Empa 10mg | Empa 25mg | Total
Number analyzed (Participants) | 165 | 165 | 168 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.6 (10.5) | 54.7 (9.9) | 54.2 (8.9) | 54.5 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 92 | 82 | 83 | 257
  Male | 73 | 83 | 85 | 241

OUTCOME MEASURES:

1. Primary Outcome: HbA1c Change From Baseline
Description: Change From Baseline in HbA1c after 24 weeks.
  Note that adjusted means are provided.
Time Frame: Baseline and 24 weeks
Population: Full analysis set (FAS) which included all randomised and treated patients who had a baseline HbA1c value. Values after start of antidiabetic rescue therapy were set to missing and last observation carried forward (LOCF) was used for imputation of missing values.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 165 | 165 | 168
percentage of HbA1c | -0.11 (0.07) | -0.59 (0.07) | -0.72 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing to adjust for multiple comparisons within each dose level, alpha split equally between the doses (2.5%). Empa versus placebo change from baseline in HbA1c was the first step in each hierarchical sequence; Based on ANCOVA with terms for treatment, background antidiabetic medication, renal function at baseline and baseline HbA1c; Mean Difference (Final Values) = -0.48, 97.5% CI 2-sided [-0.69 to -0.27], Standard Error of Mean 0.09 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.61, 97.5% CI 2-sided [-0.82 to -0.40], Standard Error of Mean 0.09 — Difference calculated as empa 25mg minus placebo

2. Secondary Outcome: Fasting Plasma Glucose (FPG) Change From Baseline
Description: Change from baseline in fasting plasma glucose (FPG) after 24 weeks of treatment.
  Note that adjusted means are provided.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: mg/dL
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 165 | 163 | 168
mg/dL | 6.47 (2.61) | -17.00 (2.63) | -21.99 (2.59)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing to adjust for multiple comparisons within each dose level, alpha split equally between the doses (2.5%). Empa versus placebo change from baseline in FPG was the second step in each hierarchical sequence; Based on ANCOVA with terms for treatment, background antidiabetic medication, renal function at baseline, baseline HbA1c and baseline FPG; Mean Difference (Final Values) = -23.48, 97.5% CI 2-sided [-31.81 to -15.15], Standard Error of Mean 3.71 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 2, analysis 1]; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -28.46, 97.5% CI 2-sided [-36.73 to -20.19], Standard Error of Mean 3.68 — Difference calculated as empa 25mg minus placebo

3. Secondary Outcome: Body Weight Change From Baseline
Description: Change from baseline in body weight after 24 weeks.
  Note that adjusted means are provided.
Time Frame: Baseline and 24 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: kg
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 165 | 165 | 168
kg | 0.34 (0.21) | -1.62 (0.21) | -1.47 (0.21)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing to adjust for multiple comparisons within each dose level, alpha split equally between the doses (2.5%). Empa versus placebo change from baseline in body weight was the third step in each hierarchical sequence; Based on ANCOVA with terms for treatment, background antidiabetic medication, renal function at baseline, baseline HbA1c and baseline weight; Mean Difference (Final Values) = -1.95, 97.5% CI 2-sided [-2.64 to -1.27], Standard Error of Mean 0.30 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 3, analysis 1]; [statistical method as in outcome 3, analysis 1]; Mean Difference (Final Values) = -1.81, 97.5% CI 2-sided [-2.49 to -1.13], Standard Error of Mean 0.30 — Difference calculated as empa 25mg minus placebo

4. Primary Outcome: HbA1c Change From Baseline for Pio and Met Background Medication Patients
Description: Change From Baseline in HbA1c after 24 weeks for patients with pioglitazone (pio) and metformin (met) background medication only.
  Note that adjusted means are provided.
Time Frame: Baseline and 24 weeks
Population: Full analysis set (FAS) which included all randomised and treated patients who had a baseline HbA1c value for patients on pioglitazone and metformin background medication. Values after start of antidiabetic rescue therapy were set to missing and last observation carried forward (LOCF) was used for imputation of missing values.
Measure: Mean (Standard Error); unit: percentage of HbA1c
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 124 | 125 | 127
percentage of HbA1c | -0.11 (0.08) | -0.55 (0.08) | -0.70 (0.07)
Statistical Analysis 1: Comparison: Placebo vs Empa 10mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — Hierarchical testing to adjust for multiple comparisons within each dose level, alpha split equally between the doses (2.5%). Empa vs placebo change from baseline in HbA1c for pio+met background only was the fourth step in each hierarchical sequence; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.45, 97.5% CI 2-sided [-0.69 to -0.21], Standard Error of Mean 0.11 — Difference calculated as empa 10mg minus placebo
Statistical Analysis 2: Comparison: Placebo vs Empa 25mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 4, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.60, 97.5% CI 2-sided [-0.83 to -0.36], Standard Error of Mean 0.11 — Difference calculated as empa 25mg minus placebo

5. Other Pre Specified Outcome: Hypoglycaemic Events
Description: Number of patients with hypoglycaemic events, as reported as adverse events.
Time Frame: From first drug administration until 7 days after last intake of study drug, up to 256 days
Population: Treated set which included all patients treated with at least one dose of randomised study medication
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Number analyzed (Participants) | 165 | 165 | 168
percentage of participants | 1.8 | 1.2 | 2.4

ADVERSE EVENTS:
Time Frame: From first dose of randomised study medication until 7 days after the last dose, up to 256 days
Arm/Group | Placebo | Empa 10mg | Empa 25mg
Serious Adverse Events (participants affected / at risk) | 7/165 | 7/165 | 6/168
Other Adverse Events (participants affected / at risk) | 56/165 | 50/165 | 34/168
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=165) | Empa 10mg (N=165) | Empa 25mg (N=168)
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1
Diabetic retinopathy (Eye disorders) | 0 | 1 | 0
Anal fissure (Gastrointestinal disorders) | 1 | 0 | 0
Constipation (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal rupture (Gastrointestinal disorders) | 0 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Amoebic colitis (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 1 | 1
Dengue fever (Infections and infestations) | 0 | 0 | 1
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 0 | 1
Urosepsis (Infections and infestations) | 0 | 1 | 0
Hand fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Brain stem infarction (Nervous system disorders) | 0 | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=165) | Empa 10mg (N=165) | Empa 25mg (N=168)
Urinary tract infection (Infections and infestations) | 18 | 24 | 18
Dyslipidaemia (Metabolism and nutrition disorders) | 17 | 18 | 12
Hyperglycaemia (Metabolism and nutrition disorders) | 26 | 8 | 4
Hypertension (Vascular disorders) | 9 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.